CLINICAL TRIAL: NCT02168322
Title: Perforated Barrier Membranes Maintain Physiologic Gingival Crevicular Fluid Growth Factor Levels During Treatment of Intrabony Defects: An In Vivo Proof-of-Principle Study
Brief Title: Perforated Barrier Membranes Maintain Physiologic Gingival Crevicular Fluid Growth Factor Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Y Gamal, professor, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Al Azhar universty
Record Dates: First submitted 2014-06-07; First posted 2014-06-20 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Vascular Endothelial Growth Factor Overexpression; Membrane Alteration
Keywords: growth factors; periodontal regeneration; modefied perforated membranes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- collagen membranes (Experimental): collagen barrier that help in isolating unwanted tissues in periodontal regneration
  Interventions: Device: collagen membrane

INTERVENTIONS:
Device: collagen membrane — bovine collagen membrane used for selective tissue regeneration
  Other Names: guided tissue membranes; guided bone regeneration; occlusive membranes
Device: collagen membrane — collagen bovine occlusive membrane for selective tissue regneration
  Other Names: guided tissue membranes; resorbable membranes; guided bone regeneration

SUMMARY:
Membrane modifecation:

Guided tissue membrane perforations may serve as a more biologic scaffold that could allow for the free passage of biologic mediators from the periosteum and overlying gingival connective tissue into the periodontal defects.

Study hyposethis:

To test this hyposthesis, this study was designed to evaluate levels of vascular endothelial cell growth factors and platlet derived growth factors in gingival crevicular fluid (GCF) during the early stages of healing for localized intrabony defects treated with modified perforated membranes (MPMs), occlusive membranes (OMs) as compared to open flap debridement control (OFD).

Methods: Thirty non-smoking patients with severe chronic periodontitis participated in this prospective, randomized and single blinded trial. Each patient contributed one interproximal defect that was randomly assigned to experimental modified perforated membrane group (10 sites), occlusive membrane group (10 sites) or open flap debridement control (10 sites). Plaque index, gingival index, probing depth (PD), clinical attachment level (CAL) and the intrabony depth of the defect (IBD) were measured at baseline for patients enrollment. Gingival crevicular fluid (GCF) samples were collected on day 1 and 3, 7, 14, 21, and 30 days after therapy. The primary outcome variable was the change in VEGF and PDGF-BB levels for sites treated by MPMs or OM compared to that of the OFD treated cases.

DETAILED DESCRIPTION:
surgical procedures:

* All surgeries were performed by the same operator (AYG).
* The surgical treatment phase was initiated only if the subject had a full-mouth dental plaque score of less than one and site plaque score of 0.
* Surgical procedures were accomplished as described in detail by Gamal and Iacono. 14 Under local anesthesia, a mucoperiosteal flap was elevated starting with an internal bevel incisions to the mucogingival junction to allow passive closure. Debridement of all inflammatory granulation tissue from the intrabony defect was performed by means of Gracey 7/8 metal curettes until a sound, healthy bone surface was obtained. At this time point, teeth were thoroughly root planed combining the use of metal curettes and power-driven instrumentation.
* For MPM treated sites, collagen membrane perforations were prepared just before surgery using a custom made 1 mm diameter pin and 1mm perforated acrylic template with a coronal occlusive rim of about 3 mm . Inter-perforation spaces were determined to be not less than 2mm in order to avoid loss of membrane stiffness. Thereafter, collagen membranes were hydrated in sterile saline, trimmed according to the template prepared for each defect, and adapted over the defects in such a manner that the entire defect and ≥2 of the surrounding alveolar bone was completely covered to avoid membrane collapse within the defect. The membranes were extended supracrestally 1 mm below the CEJ to ensure optimum gingival CT involvement in supracrestal wound healing. Collagen membranes were simply adapted in place according to the surgical protocol of the manufacturer without suturing. The mucoperiosteal flap was coronally positioned covering the entire membrane and sutured with 5-0 non-resorbable suture .
* No periodontal dressing was applied. OM and OFD sites were treated the same way except for using occlusive membranes or defect closure without using membranes. All patients received oral and written postoperative instructions.
* Patients were prescribed amoxicillin (500 mg)‡ every 8 hours for 1 week. Subjects with allergies to amoxicillin and derivatives were prescribed Clindamycin (300 mg) every 8 hours.
* Plaque control effort was supplemented by rinsing with chlorhexidine (0.12% chlorhexidine hydrochloride §) for one minute three times daily for 2 weeks. The patients were instructed to refrain from tooth brushing and interdental cleaning was avoided at the surgical areas during this time.
* Sutures were removed 14 days postoperatively and recall appointments for observation of any adverse tissue reaction and oral hygiene reinforcement were scheduled every second week during the first 2 months after surgery.
* One month after surgery, all patients were instructed to resume their normal mechanical oral hygiene measures, which consisted of brushing using a soft toothbrush with a roll-technique and flossing. Supportive periodontal maintenance including oral hygiene reinforcement and supragingival scaling was performed during each recall appointment.

Gingival Crevicular Fluid (GCF) Sampling:

To avoid irritation, samples were obtained 1 day following surgery and after individuals had fasted overnight and between 8:00AM and 10:00AM.

* Using micropipettes (5 ul), GCF samples were collected 21 by a single examiner (MA) who was masked to the attribution of the sites to groups.
* Following the isolation and drying of the selected site with cotton rolls, a fisher brand disposable micropipettes € was placed intrasulcularly at the mesiofacial line angle of the selected site to a maximum depth of 2 mm below the gingival margin. Micropipettes were left in place until 5 µl of fluid was collected.
* GCF samples were collected at day 1, 3, 7, 14, 21, and 30 days after therapy and diluted in saline solution (50 µl) for evaluation of VEGF and PDGF-BB levels. Samples were labeled, carried in a dark container and kept at -26 C until used.

ELIGIBILITY:
Inclusion Criteria:

1. no systemic diseases which could influence the outcome of the therapy;
2. good compliance with the plaque control instructions following initial therapy; 3) teeth involved were all vital with no mobility ;

4) each subject contributed a single 2 or 3-wall intrabony interproximal defects around premolar or molar teeth without furcation involvement; 5) selected 2- or 3-wall intrabony defects (IBC) measured from the alveolar crest to the defect base in diagnostic periapical radiographs of≥ 3 mm 6) selected probing depth (PD) ≥ 6 mm and clinical attachment loss (CAL) ≥ 5 mm at the site of intraosseous defects four weeks following initial cause-related therapy; 6) availability for the follow-up and maintenance program; 7) absence of periodontal treatment during the previous year; 8) absence of systemic medications that could affect healing or antibiotic treatment during the previous 6 months; and 9) absence of occlusal interferences, open interproximal contacts (diastema, flaring or both).

Exclusion Criteria:

* Pregnant females were excluded from participating in the study

Ages: 26 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
platelet derived growth factor and endothelial cell growth factor levels in the gigival cervicular fluid during Treatment of Intrabony Defects: An in Vivo Proof-of-Principle Study | 30 days
  membrane perforations could provide more physiologic growth factors concentrations in the defect area for their optimal effects. To test this assumption in a more controlled manner with a standard growth factors levels of open flap debridement treated sites, the objective of this study was to evaluate levels of platelet derived growth factors - BB (PDGF-BB) and vascular endothelial cell growth factor (VCGF) in GCF during the early stages of healing for sites treated with MPM or OM as compared with those sites treated with control OFD.

SECONDARY OUTCOMES:
clinical corelation with the growth factors levels | 30 days
  could this controled level of the growth factors acheived with perforated membrane has a clinical impact

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Y Gamal, PhD, Principal Investigator — Ain Shams Universty
Locations (1):
- Ain Shams Universty, Cairo, Nasr City, Egypt

REFERENCES:
- [Background] Gamal AY, Iacono VJ. Enhancing guided tissue regeneration of periodontal defects by using a novel perforated barrier membrane. J Periodontol. 2013 Jul;84(7):905-13. doi: 10.1902/jop.2012.120301. Epub 2012 Sep 24. PMID 23003916